CLINICAL TRIAL: NCT00744900
Title: A Phase II Trial With Pemetrexed Plus Cisplatin as First Line Chemotherapy for Advanced Non - Small Cell Lung Cancer (NSCLC) Patients With Measurable Asymptomatic Brain Metastasis (GFPC 07-01/METAL).
Brief Title: Pemetrexed Plus Cisplatin for Brain Metastasis of Advanced Non - Small Cell Lung Cancer (NSCLC)
Acronym: GFPC 07-01
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University Hospital, Brest (Other)
Responsible Party: Gilles ROBINET/MD, CHU BREST, Institut de Cancerologie et d'Hématologie
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GFPC 07-01; RB 07.103
Record Dates: First submitted 2008-08-29; First posted 2008-09-01 (Estimated); Last update posted 2009-07-28 (Estimated); Status verified 2009-07

CONDITIONS: Lung Cancer
Keywords: Pemetrexed, Non-Small Cell Lung Cancer, brain metastasis
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung; Brain Neoplasms | interventions — Pemetrexed; Cisplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- A (Experimental)
  Interventions: Drug: Pemetrexed, cisplatin

INTERVENTIONS:
Drug: Pemetrexed, cisplatin — Alimta 500mg/m² IV 10 min infusion and Cisplatin 75mg/m² IV 60 min on day 1. Cycle will be repeated each 21 days.Folic acid orally 400µg should begin 5-7days prior to the first dose of pemetrexed and continuing daily until 3 weeks after the last dose of pemetrexed. Vitamin B12 will be administered as a 1000 mg intramuscular injection, approximately one week before Day 1 of cycle 1 and should repeat approximately every 9 weeks Dexamethasone, 4 mg or equivalent, should be taken orally twice per day on the day before, the day of, and the day after each dose of pemetrexed.WBRT will be administered with high energy photons systematically after cycle 6 or in case of stable disease (SD) after cycle 4 or progressive disease (PD) at any time. The dose will be 3Gy by fraction, 1 fraction per day, for 10 days.

SUMMARY:
NSCLC patients often have cerebral metastasis : 10% at diagnosis and 40% during disease management. Neurosurgery is not indicated in the majority of cases because of presence of several lesions in the brain, failure of primary tumor control or presence of extra-cerebral metastasis. Cerebral metastasis lead to death in 30 to 50% of these cases. Management of these patients in this situation is based on supportive care and whole-brain radiotherapy. The place of chemotherapy for patients with good performance status was discussed for a long time and it is now admitted. However, the place of new drugs such as pemetrexed, which is currently used as a second line treatment for NSCLC, needs to be further studied. It is known that pemetrexed when added to cisplatin for treatment of NSCLC provides a similar effectiveness when compared to other drugs associations commonly used in this indication. In addition, Cisplatin with Pemetrexed probably present a better safety profile.

The present study is based upon the hypothesis stipulating that the association cisplatin-pemetrexed will be at least as efficient as the others association currently used for treatment of NSCLC and will present a better safety profile. The primary objective of this study is overall response rate on brain metastasis according to RECIST criteria. Secondary judgment criterias are : Overall response rate, PFS after first-line CDDP plus pemetrexed, safety profile, quality of life, neurological symptoms, overall survival.

The trial will enroll up to 45 patients in this single-arm two-stage sequential phase II study with the possibility of stopping the study early because of lack of efficacy.

ELIGIBILITY:
Inclusion Criteria:

* Patients with cytologically or histologically confirmed NSCLC.
* Patient with brain metastasis not amenable to surgery or radiosurgery with curative intent
* At least one brain measurable lesion using RECIST criteria
* ECOG Performance Status ≤2
* No prior chemotherapy for this cancer
* Prior surgery is allowed provided there is a relapse or progression after the procedure.
* Adequate organ function including the following: Adequate bone marrow reserve: absolute neutrophil count (ANC) superior or equal to 1.5 X109/L, platelets superior or equal to 100 X 109/L, and hemoglobin superior or equal to 9 g/dL; Hepatic: bilirubin <1.5 times the upper limit of normal (ULN), alkaline phosphatase (AP), aspartate transaminase (AST) and alanine transaminase (ALT) <3xULN (or <5xULN with liver metastases); Renal: Calculated creatinine clearance (CrCl) superior or equal to 45mL/min based on the standard Cockroft and Gault formula
* Signed informed consent document from the patient
* Patient must be at least 18 years of age.
* Estimated life expectancy of at least 12 weeks.
* Effective contraception (men and women) for and during the 6 months following the end of treatment

Exclusion Criteria:

* Symptomatic brain metastasis
* Have received prior radiotherapy for brain metastasis
* Unable or unwilling to take folic acid, vitamin B12 supplementation or dexamethasone (or equivalent corticosteroid); or any other inability to comply with protocol or study related procedures.
* A prior malignancy other than NSCLC, except carcinoma in situ of the cervix or non-melanoma skin cancer, adequately treated low grade [Gleason score <6] localized prostate cancer, unless that prior malignancy was diagnosed and definitively treated at least 5 years previously with no subsequent evidence of recurrence
* Serious concomitant systemic disorders (for example, active infection or abnormal electrocardiogram (ECG) indicative of cardiac disease) that, in the opinion of the investigator, would compromise the safety of the patient and his/her ability to complete study.
* Inability to discontinue administration of aspirin at a dose >1.3g/day or other non-steroidal anti-inflammatory agents for 2 days before, the day of, and 2 days after the dose of pemetrexed (5 days prior for long-acting agents such as piroxicam).
* Presence of fluid accumulations in third spaces, e.g., ascite or pleural effusion, which can be detected clinically (during physical examination), and which cannot be adequately controlled by drainage or other procedures prior to inclusion in the study.
* Peripheral neuropathy > CTC Grade 2
* Patient compliance or geographic distance precluding adequate follow up.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2008-09

PRIMARY OUTCOMES:
Objective of this study is overall response rate on brain metastasis according to RECIST criteria. | After cycles 2, 4 and 6 and every 6 weeks after study drug completion in absence of disease progression.

SECONDARY OUTCOMES:
Overall response rate, PFS after first-line CDDP plus pemetrexed, safety profile, quality of life, neurological symptoms and overall survival. | After cycles 2, 4 and 6 and every 6 weeks after study drug completion.

CONTACTS AND LOCATIONS:
Overall Officials: Gilles Robinet, MD, Principal Investigator — CHU Brest; Barlesi Barlesi, MD, Ph.D, Principal Investigator — Assistance Publique Hôpitaux de Marseille; Isabelle Monet, MD, Principal Investigator — Centre Hospitalier, Créteil
Locations (25):
- France (25):
  - Centre Hôspitalier du Pays d'Aix, Service des Maladies Respiratoires, Aix-en-Provence
  - CHU d'Angers, Service de Pneumologie, Angers
  - Médecine 4, C.H.G. de la Fontonne Antibes, Antibes
  - CHU brest, institut de cancérologie et d'hématologie, Brest
  - Centre François Baclesse, Caen
  - Centre Hospitalier René Dubos - Pontoise, Service d'Oncologie - Hématologie Clinique, Cergy-Pontoise
  - Centre Hospitalier, Service de Pneumologie, Charleville
  - CHI, Service de Pneumologie, Créteil
  - Pneumologie, Centre hôspitalier, DRAGUIGNAN, Draguignan
  - CH GAP, Gap
  - Centre Hospitalier Départemental, Service de Pneumologie,, La Roche-sur-Yon
  - Hôpital A. Mignot, Service de Pneumologie, Le Chesnay
  - Hopital de la Croix Rousse, Lyon
  - Centre Hôspitalier, Service de Pneumo-Neuro, Mantes-la-Jolie
  - Hôpital Sainte Margueritte, Marseille
  - Serv. de Pneumo-Allergo, CH de Martigues, Martigues
  - Serv. de Pneumo - Hôpital St Antoine, Paris
  - Service Pneumologie, Pavillon 1A, CH de Lyon-Sud, Pierre-Bénite
  - Hôpital Pontchailloux, Service de Pneumologie., Rennes
  - CHG, Service de Pneumologie, Roanne
  - Luc THIBERVILLE, Rouen
  - CHU de ROUEN, Hôpital Bois Guillaume, Serv. de Pneumo., Rouen
  - Institut de Cancérologie de la Loire, Saint-Priest-en-Jarez
  - CHU, Service du Pr. Carles, Toulouse
  - Pneumologie, Centre Hospitalier, Villefranche-sur-Saône